CLINICAL TRIAL: NCT05786469
Title: A Prospective, Double-blind, Randomized, Single Centre Trial to Evaluate the Rate of RAAS Inhibitor Withdrawal or Down-titration in Non-dialysis Patients with CKD Stage IIIb to V Randomized to Patiromer or Placebo (DROP)
Brief Title: Patiromer Trial in CKD Stage IIIB to V
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to reach planned study sample size due to increased patient failure to meet inclusion criteria.
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Vifor Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DROP; 2023-503984-41-00 (Other: EMA)
Record Dates: First submitted 2023-03-01; First posted 2023-03-27 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Hyperkalemia
Keywords: Chronic Kidney Diseases; Hyperkalemia; Potassium Binders
MeSH Terms: conditions — Hyperkalemia; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: DOUBLE-BLIND, RANDOMIZED, SINGLE CENTRE TRIAL
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Active study treatment and placebo will be provided by Vifor Pharma and will be indistinguishable from one another in terms of labelling and instructions.
  Allocation to one of the two treatments will be determined by the randomization's number based on a computer-generated randomization list developed by the Mario Negri Biostatistics Laboratory.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participants randomized to receive one 8.4 g packet of patiromer per day (Experimental): Patiromer is an organic, non-absorbed, sodium-free, potassium-binding polymer that exchanges potassium for calcium in the gastrointestinal tract.
  Interventions: Drug: Veltassa Oral Powder Product
- Participants randomized to receive one identical packet containing placebo (Placebo Comparator): Active study treatment and placebo will be provided by Vifor Pharma and will be indistinguishable from one another in terms of labelling and instructions
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Veltassa Oral Powder Product — The recommended starting dose is 8.4 g of patiromer, once daily (equivalent to one packet of the active ingredient, once daily). The daily dose may be adjusted in intervals of one week or longer, based on the serum potassium level and the desired target range. The daily dose may be increased or decreased by 8.4 g as necessary to reach the desired target range, up to a maximum dose of 25.2 g daily. If serum potassium falls below the desired range, the dose should be reduced or discontinued.
  Patients are expected to be included during an 18-month recruitment period. The last randomized patient will be maintained on active follow-up for 6 months. All other randomized patients will be maintained on active follow-up until the last randomized patient will have completed the planned 6-month follow-up period. Thus, the follow-up period will be expected to range from a minimum of 6 months for the last randomized patient to a maximum of 24 months for the first randomized patient
  Arms: Participants randomized to receive one 8.4 g packet of patiromer per day
Other: Placebo — The recommended starting dose is 8.4 g of patiromer, once daily (equivalent to one packet of the active ingredient, once daily). The daily dose may be adjusted in intervals of one week or longer, based on the serum potassium level and the desired target range. The daily dose may be increased or decreased by 8.4 g as necessary to reach the desired target range, up to a maximum dose of 25.2 g daily. If serum potassium falls below the desired range, the dose should be reduced or discontinued.
  Patients are expected to be included during an 18-month recruitment period. The last randomized patient will be maintained on active follow-up for 6 months. All other randomized patients will be maintained on active follow-up until the last randomized patient will have completed the planned 6-month follow-up period. Thus, the follow-up period will be expected to range from a minimum of 6 months for the last randomized patient to a maximum of 24 months for the first randomized patient
  Arms: Participants randomized to receive one identical packet containing placebo

SUMMARY:
This phase III, prospective, randomized, double-blind, placebo-controlled trial will primarily aim to compare the effects of patiromer and placebo on the rate of withdrawal or down-titration of RAAS inhibition therapy because of refractory hyperkalemia (serum K+ levels ≥ 5.5 mEq/L at two consecutive visits, one-week apart) in non-dialysis patients with CKD stage IIIB to V receiving best available conservative therapy, including RAAS inhibition with ACE inhibitors and/or ARBs and/or aldosterone antagonists. Patients are expected to be included during an 18-month recruitment period. All randomized patients will be maintained on active follow-up for 12 months. At 12 months, a final visit will be performed for all patients who complete the follow-up period. During this final visit, all the parameters evaluated at baseline will be reassessed and the study treatment will be discontinued. Whenever feasible, a final visit will be planned within one month also for those patients who prematurely discontinue the treatment period for any intercurrent reason (adverse event, consent withdrawal and other). After the final visit the patient will be discharged from the study and will be referred to his nephrologist with the suggestion to check serum potassium levels within three days.

DETAILED DESCRIPTION:
Refractory hyperkalemia is among the leading causes of initiation or chronic renal replacement therapy (RRT) by extracorporeal or peritoneal dialysis in patients with chronic kidney disease (CKD). Dialysis therapy is lifesaving but has a major impact on patients' quality of life and is terribly expensive. Thus, deferring dialysis initiation by preventing hyperkalemia would have major implications for patients and health care providers.

Among patients with CKD, glomerular filtration rate (GFR) <45 ml/min/1.73 m2, older age, coexistence of diabetes or heart failure, and inhibition of the renin angiotensin aldosterone system (RAAS) by angiotensin-converting-enzyme (ACE) inhibitors, angiotensin receptor blockers (ARBs) or aldosterone antagonists are the major risk factors for hyperkalemia. On the other hand, RAAS inhibitors - based on randomized trial results showing the superior effect of these medications compared to other antihypertensive drug classes in slowing the progression of chronic nephropathies to end-stage renal disease (ESRD) - are first-line therapy for patients with CKD, in particular for those with proteinuric nephropathies.

However, the risk of hyperkalemia is a major impediment to adequate RAAS blockade in CKD, especially when RAAS inhibitors are used in maximal doses or are combined.

Dietary counseling, correction of metabolic acidosis and treatment with loop diuretics are key components of potassium-lowering therapy in patients with CKD. Combined therapy with potassium binders, however, is often needed to prevent or treat hyperkalemia, particularly in patients with GFR <45 ml/min/1.73 m2, concomitant diabetes and/or RAAS inhibitor therapy.

A newer potassium binder, patiromer, has been approved by FDA and EMA for the treatment of hyperkalemia. Patiromer is an organic, non-absorbed, sodium-free, potassium-binding polymer that exchanges potassium for calcium in the gastrointestinal tract. Because of the remarkably good risk/benefit profile, it is conceivable that patiromer may safely improve hyperkalemia control and reduce the need of RAAS inhibition interruption or down-titration (not only of ACE inhibitors and ARBs but also of potassium sparing diuretics such as spironolactone, eplerenone and finerenone) in patients with severe CKD. In turn, this could translate into improved nephroprotection and deferred initiation of dialysis, particularly in non-dialysis patients with CKD stage IV to V. This hypothesis, however, must be tested in prospective randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study-specific procedures.
2. Age >18 years.
3. GFR <45 ml/min/1.73m2 as per CKD-EPI equation.
4. Serum potassium ≥5.0 mEq/L (in at least two consecutive evaluations, one week apart) despite dietary counseling, optimized metabolic acidosis control, diuretic therapy as needed for blood pressure control and fluid balance, and effective blood glucose control in diabetics.
5. Concomitant therapy with RAAS inhibitors (ACE inhibitors, ARBs and aldosterone antagonists, such as spironolactone and finerenone).

Exclusion Criteria:

1. Ongoing treatment with SPS before randomization (Patient eligibility could be reassessed during the screening period after at least one week from SPS therapy withdrawal)
2. Rapidly progressive kidney disease (eGFR reduction ≥ 30% over the last three months as per CKD-Epi equation) and expected risk of progression to ESKD and need of renal replacement therapy by dialysis or transplantation within six months.
3. Active systemic autoimmune diseases.
4. Concomitant treatment with steroids or any other immunosuppressive agent.
5. Hypersensitivity to the active ingredient or any of the excipients. Patients with Hereditary Fructose Intolerance.
6. Patients with or at risk of hypercalcaemia and/or hypomagnesaemia.
7. Severe/unstable heart failure with or without decreased systolic function requiring hospitalization or changes in pharmacological therapy over the last three months.
8. Refractory severe hypertension (BP >180/100 mmHg despite optimized pharmacological treatment with at least three blood pressure-lowering medications and a diuretic).
9. Positive hepatitis C antibodies, hepatitis B virus surface antigens at screening.
10. Known to have tested positive for human immunodeficiency virus.
11. Drug or alcohol abuse.
12. Female subjects who are pregnant, lactating or who intend to become pregnant before or during the study period, or within 90 days of the last dose of study treatment. Female subjects who intend to donate ova over the same time period.
13. Male subjects who intend to donate sperm during the study period or for the 90 days following the last dose of study treatment.
14. Male and female subjects in childbearing age not using a highly effective contraception method according to the 2020 CTFG Recommendations related to contraception and pregnancy testing in clinical trials (9)
15. Inability to fully understand the potential risks and benefits related to study participation.
16. Involvement in the study planning and/or conduct.
17. Participation in another clinical study with an investigational product during the last month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-11-07 (Actual)

PRIMARY OUTCOMES:
To compare the effects of patiromer and placebo on the rate of withdrawal or down-titration of RAAS inhibition therapy because of refractory hyperkalemia | 6 months
  Number of patients who withdraw or reduce RAAS inhibition therapy because of refractory hyperkalemia (serum K+ levels ≥ 5.5 mEq/L at two consecutive visits one-week apart)

SECONDARY OUTCOMES:
To compare changes in serum potassium normalization between the two treatment groups | 6 months
  Changes in Serum potassium normalization (serum K+<5.0 mEq/l considered as a dichotomous end point) for at least two consecutive visits one week apart
To compare changes in metabolic laboratory parameters between the two treatment groups | 6 months
  Changes in: serum potassium mEq/l levels considered as a continuous variable; serum calcium (mg/dl) levels; serum phosphate (mg/dl) levels; serum Magnesium (mEq/l) levels; serum intact parathyroid hormone (mg/dl) levels; serum 1,25-dihydroxyvitamin D (mg/dl) levels; 24-hour urinary calcium (mg/24h) excretion; 24-hour urinary phosphate (mg/24h) excretion; 24-hour urinary magnesium (mg/24h) excretion; Plasma renin (μU/ml) activity; serum aldosterone (ng/dl) levels; 24-hour urinary aldosterone (μg/24h) excretion; blood pH (-) levels; blood Base Excess (mmol/l) level
To compare changes in renal function parameters between the two treatment groups | 6 months
  Changes in measured GFR (mL/min) values with iohexol plasma clearance technique; 24-hour albuminuria (μg/min) excretion; 24-hour proteinuria (g/24h) excretion; 24-hour urinary albumin/creatinine (A/C) (mg/g) ratio; 24-hour urinary protein/creatinine (P/C) (mg/g) ratio; Urinary spot morning albumin/creatinine (A/C) (mg/g) ratio; Urinary spot morning protein/creatinine (P/C) (mg/g) ratio
To compare change in clinical parameters between the two treatment groups | 6 months
  Number of participants requiring renal replacement therapy because of ESRD; number of participants requiring SPS therapy
To compare events between the two treatment groups | 6 months
  Number of Fatal and non-fatal cardiovascular events; number of serious, non-serious and treatment-related adverse events
To compare costs between the two treatment groups | 6 months
  Treatment costs for the study drugs, dialysis therapy and treatment-related complications
To compare questionnaire replies between the two treatment groups | 6 months
  Quality of life as assessed using the Italian versions of validated questionnaires such as the SF-12 questionnaire.
  All items in the questionnaire apply the same response method, but with a variable and weighted score for each item.
To compare safety between the two study groups | 6 months
  Number of participant that develop hypokalemia (K+<3.5 mEq/L); Number of participant that develop hypomagnesemia (Mg++ <1.41 mg/dL); Number of participant that withdraw study treatment because of side effects

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Remuzzi, MD, Study Director — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (1):
- Centro di Ricerche Cliniche per le Malattie Rare "Aldo e Cele Daccò", Ranica, BG, Italy

IPD SHARING:
Plan to Share IPD: No